CLINICAL TRIAL: NCT00451269
Title: Multicentric Evaluation of Rapid Diagnosis Tests for the Diagnosis of Imported Malaria.
Brief Title: Evaluation of Rapid Diagnosis Tests in Imported Malaria
Acronym: TDR-PALU
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Christophe AUCAN, Department of Clinical Research of developpement
Other Study IDs: AOR 06066
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2007-03

CONDITIONS: Malaria
Keywords: Malaria; Diagnosis; RDT; pLDH; HRP2; Patients with fever and history of travel in a malaria; country
MeSH Terms: conditions — Malaria; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Rapid diagnosis test for malaria — Rapid diagnosis test for malaria

SUMMARY:
The annual number of cases of clinical malaria worldwide is estimated to be 300-500 million leading to 1.5 million deaths. Delayed care and frequent drug resistance of Plasmodium falciparum (Pf), the most frequent form of malaria, is responsible for these deaths. Each year, 5000-8000 travellers return to France with malaria, 4/5 from Africa and with Pf. Clinical features associated with a malaria crisis are poorly predictive and misdiagnosis can be easily made. Diagnosis of accurate malaria rely on microscopic examination of stained thin and thick blood films by a well trained microscopist. Few emergency wards are specialized for tropical diseases. For most of them, malaria is a rare disease and hours are lost before accurate microscopy can permit the decision

DETAILED DESCRIPTION:
The annual number of cases of clinical malaria worldwide is estimated to be 300-500 million leading to 1.5 million deaths. Delayed care and frequent drug resistance of Plasmodium falciparum (Pf), the most frequent form of malaria, is responsible for these deaths. Each year, 5000-8000 travellers return to France with malaria, 4/5 from Africa and with Pf. Clinical features associated with a malaria crisis are poorly predictive and misdiagnosis can be easily made. Diagnosis of accurate malaria rely on microscopic examination of stained thin and thick blood films by a well trained microscopist. Few emergency wards are specialized for tropical diseases. For most of them, malaria is a rare disease and hours are lost before accurate microscopy can permit the decision The rapid diagnostic tests (RDT) for malaria are designed to give a sensitive response within 15 minutes. They are based on the immunodetection of HISTIDIN rich protein 2 (HRP2) or the Pf LACTICO dehydrogenase (PfLDH), specific of Plasmodium falciparum or plasmodial LACTICO dehydrogenase (pLDH), or aldolase, specific of gender of the four species of human malaria. Recent increase of performances and availability prompted WHO to recommend their use for the diagnosis of malaria when microscopy is unavailable. In France, competence exists on the whole of the territory but expertise is usually confined to major referral centers. We intend to evaluate the performances of 4 RDT in 6 laboratories who perform the diagnosis of malaria on patients samples who returned from tourist or family or professional trips. The simultaneous detection of the plasmodial HRP2, PfLDH, aldolase and pLDH will be compared with the thick blood film as reference. Discrepant results will be analysed by PCR. The determination of the sensitivity, the specificity, the predictive positive value and the predictive negative value of the RDT is the principal objective.

ELIGIBILITY:
Inclusion Criteria:

* No refusal by patient
* Sample for malaria diagnosis

Exclusion criteria:

* Patient who do not want to participated to the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Suspected malaria
Sampling Method: Non-Probability Sample
Enrollment: 1297 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sophie MATHERON, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital BICHAT CLAUDE BERNARD, Paris, France

REFERENCES:
- [Result] Musset L, Bouchaud O, Matheron S, Massias L, Le Bras J. Clinical atovaquone-proguanil resistance of Plasmodium falciparum associated with cytochrome b codon 268 mutations. Microbes Infect. 2006 Sep;8(11):2599-604. doi: 10.1016/j.micinf.2006.07.011. Epub 2006 Aug 10. PMID 16962361